CLINICAL TRIAL: NCT00112567
Title: A Phase I/II Study of Total Body Irradiation, Thiotepa, and Fludarabine as Conditioning for Haploidentical CD34+ Purified Peripheral Blood Stem Cell Transplants
Brief Title: Total-Body Irradiation, Thiotepa, and Fludarabine in Treating Young Patients Who Are Undergoing a Donor Stem Cell Transplant for Hematologic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 1629.00; FHCRC-1629.00; CDR0000430650 (Registry Identifier: PDQ)
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: recurrent childhood acute lymphoblastic leukemia; childhood myelodysplastic syndromes; childhood acute lymphoblastic leukemia in remission; recurrent childhood acute myeloid leukemia; childhood acute myeloid leukemia in remission; secondary acute myeloid leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; childhood chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; de novo myelodysplastic syndromes; secondary myelodysplastic syndromes; previously treated myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Accelerated Phase; Blast Crisis | interventions — fludarabine phosphate; Thiotepa; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Drug: fludarabine phosphate
Drug: thiotepa
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Chemotherapy, such as fludarabine and thiotepa, and radiation therapy may destroy cancerous blood-forming cells (stem cells) in the blood and bone marrow. Giving healthy stem cells from a donor whose blood closely resembles the patient's blood will help the patient's bone marrow make new stem cells that become red blood cells, white blood cells, and platelets.

PURPOSE: This phase I/II trial is studying the side effects of total-body irradiation, fludarabine, and thiotepa and to see how well they work in treating young patients who are undergoing a donor stem cell transplant for hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety of a conditioning regimen without anti-thymocyte globulin comprising total body irradiation, thiotepa, and fludarabine followed by CD34-positive-selected haploidentical allogeneic peripheral blood stem cell transplantation in young patients with life-threatening hematologic malignancies.

Secondary

* Determine the risk for severe graft-vs-host disease in patients treated with this regimen.
* Determine the kinetics of immune reconstitution in patients treated with this regimen.
* Determine the risk for life-threatening infections in patients treated with this regimen.

OUTLINE:

* Conditioning regimen: Patients 7 years of age and under undergo total body irradiation twice daily on days -9 to -7. Patients over 7 years of age undergo total body irradiation once on day -7. All patients receive fludarabine IV once daily on days -6 to -2 and thiotepa IV over 2 hours twice on day -5.
* CD34-positive (CD34+)-selected haploidentical allogeneic peripheral blood stem cell transplantation (PBSCT): Patients undergo CD34+-selected allogeneic PBSCT on days 0 and 2.

Patients with acute lymphoblastic leukemia or CNS disease also receive methotrexate intrathecally twice before transplantation and 4 times after day 35 post-transplantation. Male patients with lymphoid malignancies undergo additional radiotherapy to the testes.

After completion of study treatment, patients are followed for at least 100 days, at 1 year, and then periodically thereafter.

PROJECTED ACCRUAL: A total of 20 patients (10 patients ≤ 7 years of age and 10 patients > 7 years of age) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of a life-threatening hematologic malignancy, including any of the following:

  * Acute leukemia advanced beyond first remission
  * Acute leukemia in first remission* with very high-risk prognostic features, including any of the following:

    * Philadelphia chromosome-positive acute lymphoblastic leukemia (ALL)
    * ALL or acute myeloid leukemia (AML) with 11q23 chromosomal abnormality
    * Hypodiploid ALL
    * Failed to achieve first remission within 1 month after induction therapy
    * Secondary AML
  * Myelodysplastic syndromes with International Prognostic Index score > 1
  * Chronic myelogenous leukemia in accelerated or blast phase NOTE: *Must be approved by PCC
* Haploidentical family donor available

  * No suitable HLA-matched related or unrelated donor available
  * No related donor mismatched for a single HLA-A, -B, -C, -DRB1, or -DQB1 antigen available

PATIENT CHARACTERISTICS:

Age

* Under 21

Performance status

* Not specified

Life expectancy

* At least 6 months

Hematopoietic

* Not specified

Hepatic

* SGPT and SGOT < 2 times upper limit of normal (ULN)*
* Bilirubin < 2 times ULN* NOTE: *Unless due to malignancy

Renal

* Not specified

Cardiovascular

* Ejection fraction ≥ 45%

Pulmonary

* DLCO ≥ 60% of predicted

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No second bone marrow transplantation, after a first regimen containing total body irradiation
* No concurrent growth factors until day 21 post-transplantation

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* See Biologic therapy

Surgery

* Not specified

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2003-04; Study Completion 2007-07

PRIMARY OUTCOMES:
Safety

SECONDARY OUTCOMES:
Risk of severe graft-versus-host disease
Kinetics of immune reconstitution
Risk of life-threatening infections

CONTACTS AND LOCATIONS:
Overall Officials: Ann E. Woolfrey, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (2):
- United States (2):
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington